CLINICAL TRIAL: NCT05838365
Title: Immediate Versus Delayed Loading of Single Posterior Zirconia Implants: A Multicenter Randomized Controlled Clinical Trial
Brief Title: Immediate Versus Delayed Loading of Single Posterior Zirconia Implants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Antonino Palazzolo, Dr. Principal Investigator, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 74/22
Record Dates: First submitted 2023-03-05; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Dental Implant Failed; Peri-implant Mucositis; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate loading zirconia implant (Experimental): Loading of zirconia dental implant within 7 days after implant placement
  Interventions: Device: Zirconia implant
- Delayed loading zirconia implant (Active Comparator): Loading of zirconia dental implants after at least 2 months of healing
  Interventions: Device: Zirconia implant

INTERVENTIONS:
Device: Zirconia implant — (Test group; within 7 days of implant placement) versus delayed (Control group; 8 weeks after implant placement)

SUMMARY:
The main aim of the present study is to investigate implant success rate after 5 years of function of immediate (Test group; within 7 days of implant placement) versus delayed (Control group; 8 weeks after implant placement) loading of two-pieces zirconia implant, placed in pristine bone without bone regeneration. Implant success rate will be defined according to Buser's criteria. Secondary endpoints: Marginal bone level (MBL) evaluation by means of standardized radiographs; Clinical evaluation of biological (e.g. Plaque Index, PI; Probing Pocket Depth, PPD, Bleeding on Probing, BOP; suppuration upon probing/palpation) and prosthetic/technical complications; Clinical evaluation of soft tissue width, keratinized tissue, marginal and interproximal soft tissue recession; Patient reported outcome measures (PROMs) by questionnaire administration:

ELIGIBILITY:
Inclusion Criteria:

* Sistemically healthy patients
* partial edentulism
* premolar position
* molar position
* Bone width and height at least 6 and 10mm, respectively.
* Keratinized tissue, at least 1 mm at implant site
* Full understanding of the proposed surgical treatments and the protocol schedule
* Full comprehension and availability to sign the informed consent form

Exclusion Criteria:

* Heavy smokers (>10 cigarettes a day)
* Serious kidney or liver diseases
* Uncontrolled diabetes
* Bisphosphonates intake
* History of radiotherapy of the head and neck
* Current antiblastic chemotherapy
* Congenital (primary) or acquired (secondary) immunodeficiency
* Pregnant women
* Connective tissue disorders

Local exclusion criteria:

* untreated stage III/IV periodontitis
* Autoimmune diseases
* oral parafunctions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Implant success rate according to Buser's criteria | 5 years
  presence of subjective complaints related to the area of treatment; recurrent infections in the peri-implant region accompanied by suppuration; mobility of the implant fixture

CONTACTS AND LOCATIONS:
Locations (1):
- San Paolo Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Primary and secondary endpoints; indicators of central tendency; evidence summary; tables; figures.